CLINICAL TRIAL: NCT06979739
Title: The Effect of Reiki and Reflexology Massage Application on Patient's Quality of Life and Pain Level in Diabetic Neuropathy Pain
Brief Title: Reiki and Reflexology Massage Diyabetik Neuropathy Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Pinar Sahin, Lecturer, Hasan Kalyoncu University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024/38
Record Dates: First submitted 2025-04-06; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Neuropathic Pain Diagnostic Questionnaire (DN4) ≥ 4
Keywords: diabetic neuropathy
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Therapeutic Touch

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1 (Experimental)
  Interventions: Behavioral: reiki
- 2 (Experimental)
  Interventions: Behavioral: refleksologia
- 3 (No Intervention)
- 4 (Experimental)
  Interventions: Behavioral: reiki and refleksologia

INTERVENTIONS:
Behavioral: reiki — 6 week reiki
  Arms: 1
Behavioral: refleksologia — 6 week refleksologia
  Arms: 2
Behavioral: reiki and refleksologia — 6 week reiki and refleksologia
  Arms: 4

SUMMARY:
Diabetes Mellitus is a chronic endocrine and metabolic disease that occurs as a result of insufficiency, absence and/or deficiency of the insulin hormone secreted from the beta cells of the pancreas, and is characterized by hyperglycemia, disorders in carbohydrate, protein and fat metabolism, capillary membrane changes and accelerated atherosclerosis, and has a high risk of morbidity and early mortality, with the development of macrovascular and microvascular complications and a high cost of care.

Diabetic neuropathy is not always painful, but 12% of all diabetic patients are affected by symptomatic painful diabetic neuropathy, the most common chronic and earliest presenting complication.

Reflexology is a special pressure technique and energy balancing system that is performed by applying pressure to reflex points with rubbing, patting and squeezing movements to ensure healing. Reflexology; It advocates that stimulating nerve points in the feet and hands with certain techniques produces electrochemical messages, which in turn stimulate the relevant organ with the help of neurons.

Feet are widely preferred for reflexology massage due to their features such as having many nerve endings, more sensitive reflexes, being easily accessible, having a large area, and the effectiveness and comfort of the application. Reflexology massage is a supportive and complementary method, not an alternative to medical treatment.

According to the Reiki principle, everything in the universe, including the human body, consists of energy in the universe, and deviations in the energy field cause diseases.

This study aims to investigate the effects of Reiki and reflexology applications on the patient's quality of life and pain level in diabetic neuropathy pain.

ELIGIBILITY:
Inclusion Criteria:

PEOPLE WITH NEUROPATHY PAIN NEUROPATHIC PAIN IS POSSIBLE MUST HAVE DIABETES Volunteering to participate in the study,

* Being able to understand and speak Turkish and not having a hearing impairment,
* Not having any diagnosed psychiatric disorder that would reduce the ability to comprehend and understand,
* Agreeing to participate in the study.
* Having no communication problems,

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2024-06-15 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Douleur Neuropathique 4 Questions-DN4 | 6 MOUNTH
visual analog scale | 6 MOUNTH
  pain

CONTACTS AND LOCATIONS:
Overall Officials: PINAR ŞAHİN, Principal Investigator — www.hku.edu.tr; nermin olgun, Study Director — www.hku.edu.tr
Locations (2):
- Turkey (Türkiye) (2):
  - Adana City Hospital, Adana, Adana
  - Adana Hospital, Adana, Adana

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- Available data/document: Informed Consent Form — https://www.hku.edu.tr/iletisim/